CLINICAL TRIAL: NCT06713226
Title: Prospective, Multi-center, Pre-market, Assessor-blinded Study to Evaluate the Clinical Performance of the Hativ P30 Electrocardiogram Recorder Device
Brief Title: Clinical Performance Evaluation of the Hativ P30
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VUNO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: VN-P30-01
Record Dates: First submitted 2024-11-22; First posted 2024-12-03 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this study, the annotators perform labeling on the Hativ P30 and the 12-lead ECG comparator for quantitative and qualitative assessment. At that time, the annotators are blinded to which device is the Hativ P30 or the 12-lead ECG comparator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Hativ P30 and 12-lead ECG comparator device — The purpose of this study is to compare the clinical equivalence and diagnostic ability of the Hativ P30 against the 12-lead ECG comparator device.
  Electrocardiograms of all participants will be obtained using both the Hativ P30 and a 12-lead ECG comparator. That is, all participants will get the same intervention.

SUMMARY:
Hativ P30 is intended to record, store, and transfer one-and two-channel ECG rhythms, and analyze them based on an artificial intelligence (AI) algorithm. In single channel mode, Hativ P30 can record lead-I. In two-channel mode, Hativ P30 can record lead-I and lead-II simultaneously and derive Lead-III and unipolar limb leads aVR, aVF and aVL. The ECG signal measured through the device's electrode is converted into a digital signal and transmitted via Bluetooth to an Android or iOS-based smart device with a mobile app installed. The ECG signal and analysis result can be checked through the screen of the smart device.

The aim of this clinical study is to assess the safety and efficacy of the Hativ P30 ECG recording device, as well as to gather data to support an FDA submission through the 510(k) process for the device's commercialization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older
* Able to provide written informed consent
* Able to remain in the same position for an ECG recording for at least 20 minutes using a standard 12-lead ECG recorder and the Hativ P30 device
* NSR cohort only: no history of arrhythmia
* NSR cohort only: no history of cardiovascular diseases, including but not limited to hypertension, hyperlipidemia, coronary artery disease, heart failure, peripheral artery disease, and stroke
* NSR cohort only: being in NSR at the time of screening ECG
* Arrhythmia cohort only: documented persistent, permanent, or chronic arrhythmia (AF or flutter, sinus rhythm with APB, sinus rhythm with VPB)
* Arrhythmia cohort only: being in arrhythmia (AF or flutter, sinus rhythm with APB, sinus rhythm with VPB) at the time of screening ECG

Exclusion Criteria:

* Subjects with an implantable pacemaker device, implantable cardioverter-defibrillator device, or internal simulator that would generate internal interference with the recording of the Hativ P30 device or a standard 12-lead ECG recorder
* Any medical or cognitive condition that would interfere with the consenting process and study-related procedures as determined by the Investigator
* Any known clinical condition (e.g., body tremors, non-healed chest wound, limb absence, etc.) that would preclude appropriate placement of the leads and/or compromise study measurements in the opinion of the Investigator
* Poor 12-lead screening ECG quality
* Pregnant at the time of enrollment
* Participation in other interventional clinical studies that includes active treatment for the last three (3) months (observational studies and long-term follow-up [no active treatment] will be allowed)
* Screening ECG record resulting in a significant arrhythmia out of the scope of the study, such as Supraventricular Tachycardia, Ventricular Tachycardia, Ventricular Fibrillation, Neurocardiogenic Syncope, among others

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 126 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2025-07-23 (Estimated); Study Completion 2025-07-23 (Estimated)

PRIMARY OUTCOMES:
Quantitative assessment and comparison of the two devices | 30 seconds
  Median beat cross correlation for Lead I and II.
Quantitative assessment and comparison of the two devices | 30 seconds
  QRS amplitude of the median beats of all six limb leads by RMS error.
Qualitative assessment and comparison of the two devices | 30 seconds
  Diagnostic equivalence between Hativ P30 and 12-lead ECG by three cardiologists (NSR, AF or flutter, sinus rhythm with APB, sinus rhythm with VPB).

IPD SHARING:
Plan to Share IPD: No